CLINICAL TRIAL: NCT02647645
Title: Cognitive Training With and Without tDCS to Improve Cognition in HIV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pilot study protocol terminated to begin expanded study.
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1203142F
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: HIV; Mild Neurocognitive Disorder
MeSH Terms: conditions — Neurocognitive Disorders | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Training (Active Comparator): Cognitive training Sham tDCS
  Interventions: Procedure: Cognitive training; Device: Sham transcranial direct current stimulation
- Cognitive Training with tDCS (Experimental): Cognitive training Active tDCS
  Interventions: Device: Transcranial direct current stimulation; Procedure: Cognitive training

INTERVENTIONS:
Device: Transcranial direct current stimulation — Direct current stimulation at a current of 1.5 mA with anode at F3 (left dorsolateral prefrontal cortex) and cathode at Fp2 (right frontal pole) for a period of 20 minutes each for 6 sessions over two weeks simultaneously with cognitive training.
  Other Names: tDCS; Transcranial electric stimulation
  Arms: Cognitive Training with tDCS
Procedure: Cognitive training — Computer delivered intervention designed to improve cognitive speed and executive functioning for a period of 20 minutes each for 6 sessions over two weeks.
  Other Names: Brain training
Device: Sham transcranial direct current stimulation — Direct current stimulation at a current of 1.5 mA with anode at F3 (left dorsolateral prefrontal cortex) and cathode at Fp2 (right frontal pole) for a period of one minute to simulate active treatment applied in 6 sessions over two weeks.
  Other Names: Sham tDCS; Sham transcranial electric stimulation
  Arms: Cognitive Training

SUMMARY:
The purpose of this study is to develop pilot data on the potential efficacy of computer-based cognitive training or the combination of computer-based cognitive training with transcranial direct current stimulation (tDCS) in improving cognitive function in persons with HIV-related mild neurocognitive disorder (MND).

DETAILED DESCRIPTION:
The purpose of this study is to develop pilot data on the potential efficacy of computer-based cognitive training or the combination of computer-based cognitive training with transcranial direct current stimulation (tDCS) in improving cognitive function in persons with HIV-related mild neurocognitive disorder (MND). tDCS is a noninvasive brain stimulation technique in which a small direct current (1-2 mA) is applied to the scalp during a cognitive or motor activity, inducing a very small current that affects specific neural circuits related to the site at which electrodes are placed. tDCS has been judged safe and has shown significant treatment effects in studies with other populations, but has not been extensively studied in individuals with HIV infection. tDCS has been shown to facilitate learning in a number of studies, suggesting that it may improve or enhance learning in those with cognitive problems. As HIV infection is associated with decrements in a number of cognitive skills, including working memory, executive functions, and psychomotor speed that are related to individuals' functional status and medication adherence, the demonstration of a technique to enhance the effects of cognitive training in this population would have substantial clinical benefits as well as scientific value.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Fluent in English
* Meets Frascati criteria for mild neurocognitive disorder

Exclusion Criteria:

* Left handed
* Presence of dementia
* Use of specific psychotropic medications including antidepressants, antipsychotics, and sleep-promoting medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond L Ownby, MD, PhD, Principal Investigator — Nova Southeastern University
Locations (1):
- NSU Psychiatry Research Office, Fort Lauderdale, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Training: Cognitive training Sham tDCS
  Transcranial direct current stimulation: Direct current stimulation
- Cognitive Training With tDCS: Cognitive training Active tDCS
  Transcranial direct current stimulation: Direct current stimulation
Period: Overall Study
Arm/Group | Cognitive Training | Cognitive Training With tDCS
Started | 11 | 10
Completed | 9 | 9
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Training | Cognitive Training With tDCS | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.45 (10.16) | 48.70 (7.04) | 47.52 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 7
  Male | 4 | 10 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Working Memory: Participants' Rate of Improvement
Description: Participants' rate of improvement on a verbal working memory task. Participants completed a battery of cognitive measures administered by an evaluator blind to treatment assignment. We used the Digits Backward trial of the Digit Span subtest of the Wechsler Adult Intelligence Scale Fourth Edition (WAIS-IV; Pearson Assessment) to measure working memory. We used raw scores for analyses. These are the largest number of digits the participant could remember and repeat in reverse order. Possible range of scores is from zero to 10. Normal persons typically remember from 5 to 7 digits. Higher scores are considered better. Analysis results are overall estimated marginal means from repeated measures analysis of covariance with treatment group as a fixed factor and age, gender, race, education, helper T cell count, and log viral load as covariates.
Time Frame: 3 weeks
Population: All participants who completed treatment.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Training | Cognitive Training With tDCS
Number analyzed (Participants) | 9 | 9
units on a scale | 6.61 (0.62) | 7.45 (0.62)
Statistical Analysis 1: Comparison: Cognitive Training vs Cognitive Training With tDCS; Analysis results are overall estimated marginal means from repeated measures analysis of covariance with treatment group as a fixed factor and age, gender, race, education, cluster of differentiation (CD4) cell count, and log viral load as covariates; Test type: Superiority — Power calculation was based on similar studies of cognitive training with transcranial direct current stimulation (tDCS); p = 0.02, ANCOVA — Probability associated with the test of the interaction between participants' performance and session number in repeated measures analysis of covariance. In light of small sample size, estimated effect size was also calculated (d = 1.78); Test was adjusted for age, gender, race, education, CD4 count, and log viral load

2. Secondary Outcome: Center for Epidemiological Studies Depression Scale (CES-D)
Description: Participants' mood over the course of the study. We used the Center for Epidemiological Studies--Depression scale (CES-D) to measure mood. This measure includes 20 items that ask the person assessed to report his or her experience of mood symptoms over the past two weeks. Participants completed this measure before and after the study intervention. Scores can range from zero to 60, with most persons attaining a score of 15 or less. Higher scores are considered worse as they indicate more frequent or more severe mood symptoms.
Time Frame: 3 weeks
Population: All participants who completed the study.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Training | Cognitive Training With tDCS
Number analyzed (Participants) | 9 | 9
units on a scale | 12.95 (6.21) | 23.37 (5.10)
Statistical Analysis 1: Comparison: Cognitive Training vs Cognitive Training With tDCS; Results are overall estimated marginal means from repeated measures analysis of covariance with treatment group as a fixed factor and age, gender, race, education, CD4 count, and log viral load as covariates; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.34, ANCOVA — Probability associated with the test of the interaction between participants' performance and session number in repeated measures analysis of covariance. In light of small sample size, estimated effect size was also calculated (d = .71); Test was adjusted for age, gender, race, education, CD4 count, and log viral load

3. Secondary Outcome: Patient's Own Assessment of Function (PAOF)
Description: Patient report of cognitive difficulties on the Patient Assessment of Own Functioning. This scale comprises 33 items describing problems in thinking, language, and memory. Participants rate each items according to how often they experience each problem on a six-point scale from "almost never" (score of 0) to "almost always" (score of 5). The participant's score is the sum of ratings on all items. The range of possible scores on each item is from 0 to 5, with most persons achieving a score of 1.5 or lower. Higher scores represent more frequent report of cognitive difficulties and thus are considered worse. The range of all possible scores for the full scale of 33 items is is 0 to 165.
Time Frame: 3 weeks
Population: All participants who completed training.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Cognitive Training | Cognitive Training With tDCS
Number analyzed (Participants) | 9 | 9
Score on a scale | 7.39 (0.73) | 9.17 (0.73)
Statistical Analysis 1: Comparison: Cognitive Training vs Cognitive Training With tDCS; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Power calculation was based on the investigators' estimate of the impact of cognitive training with transcranial direct current stimulation (tDCS) on subjective cognitive problems, as similar studies were not available to develop effect size estimates; p = 0.33, ANCOVA — Probability associated with the test of the interaction between participants' performance and session number in repeated measures analysis of covariance. In light of small sample size, estimated effect size was also calculated (d = .63); Test was adjusted for age, gender, race, education, CD4 count, and log viral load

ADVERSE EVENTS:
Time Frame: 1 year, 3 months
Arm/Group | Cognitive Training | Cognitive Training With tDCS
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
Analyses were based on a small sample size. The sample size was smaller than originally planned, as the study was stopped when external funding for a more extensive and better controlled study was obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-12-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT02647645/Prot_000.pdf
  • Statistical Analysis Plan (2014-12-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT02647645/SAP_001.pdf